CLINICAL TRIAL: NCT04855500
Title: A Registry of Coronary Artery Optical Coherence Tomography of Hainan General Hospital
Brief Title: A Single Center Registry of Coronary OCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hainan People's Hospital (Other)
Responsible Party: Principal Investigator, Liao Wang, Deputy director of Cardiology, Hainan People's Hospital
Other Study IDs: WangLiao002
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease; Optical Coherence Tomography; Registry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry started January 1,2020 to collect patients who recieve coronary OCT imaging in Hainan General Hospital.All enrolled patients will receive 1 year followed-up.

DETAILED DESCRIPTION:
This registry started January 1,2020.Patients >= 18 years old who recieve coronary OCT imaging in Hainan General Hospital are included in current registry.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who recieved intracoronary OCT imaging during cardiac catheterization are eligible for this registry.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who recieved intracoronary OCT imaging during cardiac catheterization are eligible for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hainan General Hospital, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: Undecided